天津市糖尿病视网膜病变社区筛查研究

Community screening study of diabetic retinopathy in Tianjin

李筱荣

眼底外科

版本号及日期:

01, 2024.01.26

# 一、研究背景及立项依据

随着糖尿病在全世界范围的大流行,糖尿病视网膜病变(diabetic retinopathy, DR)作为糖尿病最常见的微血管并发症之一,已经成为造成全世界劳动年龄人口不可逆性失明的主要原因。在中国,45岁及以上的成年人 DR 的患病率为 18.45%(1316万人),世界范围内约为 34.6%(9300万人)。DR 患者约占糖尿病人群的 1/4~1/3。DR 已经成为一个严重的公共卫生问题。DR 的致盲特点属于"可防不可治",DR 早期筛查可极大降低 DR 的致盲率以及有效降低 DR 的医疗成本,因此 DR 的早期筛查显得尤为重要。早期筛查可以及时了解患者眼底情况,根据病变状态给出合适的干预措施。早期筛查和及时干预可使糖尿病患者视力丧失的风险降低 50%~70%,此外,早期筛查的成本效益比也是最优的。因此,DR 筛查工作迫在眉睫。

我们希望通过此研究了解天津市糖尿病视网膜病变的患病率及其影响因素,提升 基层医疗卫生机构糖尿病患者并发症发现干预能力,构建上下联动的糖尿病防治网络; 广泛开展宣传教育,提升患者自我管理意识,提高糖尿病视网膜病变筛查率,降低致 盲率。

# 二、研究目的

- 1. 发挥市级医院技术优势,提升基层医疗卫生机构糖尿病患者并发症发现干预能力,构建上下联动的糖尿病防治网络。
  - 2. 坚持预防为主、防治结合的工作方针,探索适宜我市的糖尿病防控模式。
- 3. 广泛开展宣传教育,提升患者自我管理意识,提高糖尿病视网膜病变筛查率, 降低致盲率。

# 三、研究设计

#### 3.1 研究现场及研究人群

在我市河西、河北、和平及滨海新区开展糖尿病视网膜病变筛查工作,每年对18000 名糖尿病患者进行眼底检查。

#### 3.2 调查内容

3.2.1确定项目承担单位

河西、河北、和平及滨海新区卫生健康委结合辖区实际,确定承担项目的基层医

疗卫生机构。基层医疗卫生机构结合基本公共卫生服务糖尿病患者管理项目,将部分 在管糖尿病患者纳入筛查项目。

#### 3.2.2 组织动员和健康教育

河西、河北、和平及滨海新区卫生健康委组织基层医疗卫生机构,做好目标人群 的宣传动员和糖尿病视网膜病变等并发症防治知识宣传,组织目标人群填写《知情同 意书》,确保筛查对象知情同意。天津医科大学眼科医院负责做好技术指导。

## 3.2.3 现场筛查

天津医科大学眼科医院、项目所在基层医疗卫生机构负责组建筛查队伍,对糖尿病患者进行眼底检查,相关检查包括视力、电脑验光、眼底照相和光相干断层扫描血管造影(OCTA)等。河西区及和平区纳入筛查患者抽血取样检测糖化血红蛋白,天津医科大学朱宪彝纪念医院负责检测糖化白蛋白和尿 ACR、四肢血管彩色多普勒超声(筛查糖尿病足风险)和中医四诊合参检查等相关指标。检查完成后对筛查人员建立健康档案。

#### 3.2.4 随访干预

对所有筛查干预对象按照风险因素分级后,针对不同级别危险人群开展有针对性的 的简 访干预工作。

- 1. 基层医疗卫生机构,对无糖尿病视网膜病变的患者建议定期随访。
- 2. 有糖尿病视网膜病变的患者,建议其转诊到上一级医疗机构进行进一步诊疗。

#### 3.3 数据管理与统计分析方案

- 3.1病例报告表/电子数据记录
- 3.2数据管理
- (1) 选择数据库excel
- (2) 建立数据库的基本框架并进行测试
- (3) 病例报告表录入前的核查以及录入人员的培训
- (4) 进行数据双录
- (5) 数据校对
- (6) 数据库锁库
- (7) 对数据库数据进行统计分析

#### 3.4 偏倚的控制

3.4.1 无应答偏倚

无应答偏倚是指由于各种原因造成没有能够获取入组观察对象的相关信息所产生的偏移。

#### 控制方法:

- 1) 科学组织调查工作,加强对调查人员的培训,在调查工作开始前最大限度地预见和解决可能造成无应答的问题。
- 2) 多次访问。实践证明调整访问策略再次或多次对调查对象进行追踪是提高应答率的一种十分有效的方法。多次访问不仅可以提高应答率,同时维护了信息的完整性。
  - 3.4.2信息偏倚

信息偏倚是指在研究实施阶段从研究对象获取信息时所产生的系统误差,主要来自于以下三个方面:

- 1)来自调查员的偏移,控制方法:加强培训、考核、检查和监督。
- 2)调查对象应答引起的偏移,控制方法:消除被调查者的顾虑,明示保护个人隐私是我们工作中最基本的职业道德。
- 3)测量偏移,控制方法:对设备条件和方法统一标准化并定期校验技术人员统一培训规范操作流程。

#### 3.5质量管理

3.5.1 职责分工

市卫生健康委负责全市项目工作的组织领导和督导检查工作。

天津医科大学眼科医院负责项目的具体实施管理、技术支持、宣传动员、评估总结、质量控制等工作,要加强数据分析,通过比较成本及产出,做好筛查项目的社会经济学评价。天津医科大学朱宪彝纪念医院负责评估红细胞寿命对于糖尿病视网膜病变进展的意义。

项目区卫生健康委负责制定辖区项目实施方案并具体组织落实,建立市级医院和各基层医疗卫生机构协作机制,做好项目日常管理工作。

基层医疗卫生机构在市级医院的指导下,采集患者的基础信息、问卷调查及常规血生化检测指标,配合做好糖尿病患者的视网膜病变筛查工作,对无风险患者开展随

访干预。

为避免给患者重复检查带来不必要的损害,对于本项目中所需数据若基层医疗卫生机构已存在或已完成采集的部分,可将数据与本项目组进行共享。

# 3.5.2项目培训

由项目地区卫生健康委牵头,天津医科大学眼科医院组织,培训对象为基层医疗卫生机构参加筛查及随访的医务人员。

## 3.5.3 经费管理

项目经费由中央转移支付重大传染病防控经费保障。各项目承担单位要设专人负责管理项目资金,专款专用。对管理不善、控制不严或违反规定弄虚作假,骗取、截留、挪用项目资金的,按照有关规定处理。

## 3.6 伦理审查与知情同意

此方案由天津医科大学眼科医院伦理委员会审批同意。筛查人员自愿签署知情同意书,可以选择不参加本项研究,或者在任何时候通知研究者要求退出研究,数据将不纳入研究结果,医疗待遇与权益不会因此而受到影响。

研究者:

年 月 日